CLINICAL TRIAL: NCT00674102
Title: An Open-label, Phase I Trial of Intravenous ASA404 Administered in Combination With Paclitaxel and Carboplatin in Japanese Patients With NSCLC
Brief Title: An Open-label, Phase I Trial of Intravenous ASA404 Administered in Combination With Paclitaxel and Carboplatin in Japanese Patients With Non-Small Cell Lung Cancer (NSCLC)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CASA404A1101
Record Dates: First submitted 2008-05-05; First posted 2008-05-07 (Estimated); Last update posted 2020-12-09 (Actual); Status verified 2016-04

CONDITIONS: Non-small Cell Lung Cancer
Keywords: Vascular disrupting agent; Non-small cell lung cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — vadimezan

ARMS (1):
- ASA404 (Experimental)
  Interventions: Drug: ASA404

INTERVENTIONS:
Drug: ASA404

SUMMARY:
The safety, tolerability, efficacy and pharmacokinetics of ASA404 when administered in combination with paclitaxel and Carboplatin are assessed. ASA404 is administered intravenously every 21 days to Japanese patients with Non small cell lung cancer.

ELIGIBILITY:
Inclusion criteria:

1. Histologically or cytologically confirmed non-small cell carcinoma of the lung.
2. Newly diagnosed Stage IIIb disease or Stage IV disease
3. No prior treatment for Stage IIIb/IV non-small cell carcinoma of the lung (Note: Prior neoadjuvant or adjuvant chemotherapy within 6 months is allowed.)
4. Age ≥ 20 years old
5. WHO Performance status of 0-1
6. Lab values within the range as defined below within 2 weeks of study registration (Note: without the use of growth factors or blood transfusions):

   * Absolute neutrophil count (ANC) > 2.0 x 109/L
   * Platelets ≥ 100 x109/L
   * Hemoglobin ≥ 9.5 g/dL
   * Serum creatinine ≤ 1.5 x ULN or 1.5 mg/dL
   * Serum bilirubin ≤ 1.5 x ULN
   * Aspartate transaminase (AST) and alanine transaminase (ALT)

     ≤ 2.5 x ULN
   * PT-INR ≤ 1.5 x ULN
   * Potassium ≥ LLN or correctable with supplements.
   * Total calcium (corrected for serum albumin) ≥ LLN or correctable with supplements.
   * Magnesium ≥ LLN or correctable with supplements.
   * Females of child-bearing potential must have negative pregnancy test (serum)
7. Life expectancy ≥ 12 weeks
8. Written informed consent obtained according to local guidelines

Exclusion criteria:

1. Patients having symptomatic CNS metastases and requiring treatment
2. Patients with second primary cancer, with the exception of non-melanoma skin cancer or cervical cancer in situ.
3. Radiotherapy ≤ 4 weeks prior to registration (In case of palliative radiotherapy 2 weeks prior to registration
4. Major surgery ≤ 4 weeks prior to registration (major surgery is defined by the use of general anesthesia). Minor surgery ≤ 2 weeks prior to registration. Insertion of a vascular access device is allowed. Patients must have recovered from all surgery-related complications.
5. Concurrent use of other investigational agents and patients who have received investigational agents ≤ 4 weeks prior to registration
6. Prior exposure to VDAs or other vascular targeting agents (anti-VEGF, anti-VEGF receptor agents, anti-EGFR agents
7. Patients with pleural effusion to be drained (Patients who have recurrence of pleural effusion and/or it takes 2 weeks before registration after drainage are allowed)
8. Patients with recent hemoptysis associated with NSCLC (>1 teaspoon in a single episode within 4 weeks)
9. Known allergy or hypersensitivity to platinum-containing drugs, taxanes, other drugs formulated in Cremophor EL (polyoxyethylated castor oil) or any known excipients of these drugs.
10. Peripheral sensory neuropathy with functional impairment (CTC Grade 2 neuropathy, regardless of causality)
11. ≥ CTC Grade 2 cardiac arrhythmias (i.e. symptomatic, but may not require medications).
12. Pregnant or breast feeding females
13. Patients who take medicine that are known to prolong the QT interval
14. Women of child bearing potential or sexually active males, unwilling or unable to use the required highly effective method(s) of contraception for both sexes while receiving treatment and for at least 6 months after the discontinuation of study treatment. (Adequate forms of contraception include IUD, oral or depot contraceptive or the barrier method plus spermicide.)
15. Patients with any one of the following

    * Patients with Long QT Syndrome
    * Patients with a Baseline 12-lead ECG QTc of > 450 msec in males or > 470 msec in females.
    * Congestive heart failure(NY Heart Association class III or IV)
    * Patients with a myocardial infarction within 12 months of study entry
    * Unstable or poorly controlled angina pectoris
    * History of poorly controlled hypertension with anti-hypertensive regimen
    * History of a sustained ventricular tachycardia
    * Any history of ventricular fibrillation or Torsades de Pointes
    * Right bundle branch block and left anterior hemiblock (bifasicular block)
    * Bradycardia defined as heart rate < 50 beat per minutes
16. Concurrent severe and/or uncontrolled medical disease (i.e. uncontrolled diabetes, chronic renal disease, chronic liver disease, confirmed diagnosis of HIV infection or active uncontrolled infection).
17. Patients known to be HBV or HCV positive
18. Significant neurological or psychiatric disorder which could compromise participation in the study
19. Patient unwilling or unable to comply with the protocol
20. Patients who are not adequate to enter the study decided by the investigator from the medical point of view.

Other protocol-defined inclusion/exclusion criteria may apply.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2008-04; Primary Completion 2009-03 (Actual)

PRIMARY OUTCOMES:
To assess the safety profile and tolerability of ASA404 when administered in combination with paclitaxel and carboplatin in Japanese patients with non small cell lung cancer | First cycle

SECONDARY OUTCOMES:
To characterize the pharmacokinetics profile of ASA404 in Japanese patients | every 2 cycles

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (4):
- Japan (4):
  - Novartis Investigative Site, Aichi
  - Novartis Investigative Site, Osaka
  - Novartis Investigative Site, Shizuoka
  - Novartis Investigative Site, Tokyo

REFERENCES:
- See also: Results for CASA404A1101 can be found on the Novartis Clinical Trial Results Website — https://www.novctrd.com/ctrdweb/trialresult/trialresults/pdf?trialResultId=3520